CLINICAL TRIAL: NCT00761059
Title: Prospective, Placebo-Controlled Blinded Clinical Trial to Study the Efficacy of Orally Administered Glucose 20% for Relieving Pain During Nasopharyngeal Suctioning in Preterm Infants > 1500g Under CPAP-Therapy
Brief Title: Analgesic Efficacy of Oral Glucose in Preterm Neonates During Suctioning
Acronym: Glucose FG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Dr. med Christoph Huenseler, University of Cologne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Uni-Koeln-905
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Analgesia
Keywords: analgesia; infant, premature; glucose; nasopharyngeal suctioning
MeSH Terms: conditions — Agnosia; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose 20% (Active Comparator)
  Interventions: Drug: Glucose 20%
- placebo (Placebo Comparator)
  Interventions: Drug: Aqua

INTERVENTIONS:
Drug: Glucose 20% — The oral application of 0,3 ml/kg Glucose 20% 3 minutes before nasopharyngeal suctioning
  Arms: Glucose 20%
Drug: Aqua — The oral application of 0,3 ml/kg Aqua 3 minutes before nasopharyngeal suctioning
  Arms: placebo

SUMMARY:
Nasopharyngeal suctioning is a painful procedure that often becomes necessary in the care of preterm infants under CPAP therapy several times a day. Since the use of analgetic and sedative drugs is accompanied with multiple side effects these are usually being avoided. Glucose 20% has been shown to have an analgesic effect when administered to preterm infants previous to some painful procedures (i.e blood sampling).

In this clinical trial the efficacy of orally administered Glucose 20% for relieving the procedural pain of nasopharyngeal suctioning is tested. The investigators' study has a cross-over design and is to include 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns (>1500g birth weight) up to a gestational age of 36+6 weeks
* CPAP respiratory therapy
* Parents' given written consent

Exclusion Criteria:

* Diseases complicating neuromuscular evaluation.
* Drug abuse by the mother
* Administration of other analgetic or sedative drugs within the previous 48h.
* Participation in another interventional clinical trial within 4 weeks before the beginning of this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The PIPP-Score, a validated pain-score, is used to measure the patient's pain | during nasopharyngeal suctioning

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Huenseler, Dr med, Principal Investigator — Neonatology, Children's Hospital, University of Cologne
Locations (1):
- Neonatology, Children's Hospital, University of Cologne, Cologne, Germany